CLINICAL TRIAL: NCT06895213
Title: Evaluation of Plasma Renin Concentrations in Cardiac Surgery
Status: Recruiting | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Patrick M. Wieruszewski, Pharm.D., Assistant Professor of Anesthesiology, Mayo Clinic
Other Study IDs: 24-004256
Record Dates: First submitted 2025-03-13; First posted 2025-03-26 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-05

CONDITIONS: Cardiac Surgery With Cardiopulmonary Bypass
Keywords: renin-angiotensin system; RAS; hypotension; perfusion; shock; blood pressure
MeSH Terms: conditions — Hypotension; Shock

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this research is to learn more about how renin (a blood test) is affected by cardiopulmonary bypass, the heart-lung machine used during open heart surgery. Renin is a protein that may be elevated in response to low blood pressure or situations where organs do not receive sufficient oxygen. Renin may potentially be used as an indicator for specific treatments aimed to increase the blood pressure. This study will evaluate blood samples for renin concentration throughout the course of open heart surgery.

DETAILED DESCRIPTION:
The investigator hypothesizes that renin concentrations will increase with exposure to cardiopulmonary bypass and that increased renin concentrations will be associated with the development of vasoplegia.

Specific Aim 1. To characterize the effects of cardiopulmonary bypass on plasma renin concentrations in adults undergoing cardiac surgery.

Specific Aim 2. To test the prognostic value of plasma renin concentrations on outcomes following cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

* Adult persons 18 years of age or greater.
* Scheduled for an elective cardiac surgical procedure involving the use of cardiopulmonary bypass.

Exclusion Criteria:

* Surgery involving heart or lung transplantation or implant of a durable left ventricular assist device.
* Emergency cardiac surgery.
* Established diagnosis of any congenital heart disease.
* End-stage kidney disease receiving kidney replacement therapy before surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult persons 18 years of age or greater (female and male).
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-04-14 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Plasma renin concentrations | Up to 24 hours after surgery

SECONDARY OUTCOMES:
Vasoplegia | First 24 hours postoperative
  Requirement of any vasopressor to maintain a mean arterial pressure of 65 mmHg or greater despite a cardiac index of at least 2.2 L/min/m2 with or without the need for pharmacologic inotropy
Acute kidney injury | 7 days
  Assessed by the Kidney Disease Improving Global Outcomes (KDIGO) staging criteria
Organ dysfunction | 28 days
  The presence of any organ support therapy including vasopressors, renal replacement therapy, and mechanical ventilation
Mortality | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Patrick M Wieruszewski, Pharm.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No